CLINICAL TRIAL: NCT00319085
Title: Comparison Between Preheated and Non-preheated Femur Component in Hybrid Total Hip Arthroplasty (THA) A Prospective Randomized Study of the 80 THA Using Radiostereometry.
Brief Title: Preheating of Femur Component in Hybrid Total Hip Arthroplasty
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Northern Orthopaedic Division, Denmark (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ON-04-008a-JPE
Record Dates: First submitted 2006-04-27; First posted 2006-04-27 (Estimated); Last update posted 2015-04-10 (Estimated); Status verified 2015-04

CONDITIONS: Osteoarthritis, Hip
Keywords: Arthroplasty,; Hip,; Pre-heating,; Radiostereometric analysis,; Dual-Energy Radiographic Absorptiometry,
MeSH Terms: conditions — Osteoarthritis, Hip | interventions — Arthroplasty, Replacement, Hip

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Procedure: Total hip replacement (Preheating of femur stem) — Total hybrid hip arthroplasty, cementation of femural component, preheating, radiostereometry, DEXA

SUMMARY:
Background

* Recently published studies confirm that preheating of femoral component enhances shear strength of implant-cement interface. Both Iesaka et al 2003 and Jafri et al 2004 showed reduction in cement porosity on cement-implant interface with preheated femur components. We will use the radiostereometry analysis (RSA) to investigate how the preheating of femur component influence on prosthesis survivorship. There are no clinical controlled studies performed to the date.

The aim of the study

* Comparison of the migration rates between preheated and non-preheated femur components, analyzed with RSA.

Methods

* Randomization of 80 patients into 2 groups with 40 in each. All patients will undergo standard hybrid total hip replacement. In group one the femur component (Bi-Metric, Interlock Biomet) will be preheated to 40 degrees of Celsius before cementation. In group two: the control group, the femur component will be of room temperature. We will measure the temperature at cement bone interface during the operation with use of thermocouple electrodes inserted through separate drill hole in the femur. The measurements will be recorded every 10 seconds. The patients will follow the standard postoperative rehabilitation program.
* The RSA analysis will be performed the first day after the operation and at 3, 12, 24 months postoperatively.
* The Dual-energy X-ray absorptiometry scanning (DEXA) of the femur will be performed at the first week after the operation and at 12 and 24 months postoperatively.
* The patients will be followed both clinically and radiologically at 1 and 2 years after the operation (Harris Hip Score).
* The results will be expressed as mean + SD (in mm). ANOVA statistical analysis will be used to confirm the differences between the groups.

ELIGIBILITY:
Inclusion Criteria:

* The patients suffering of hip osteoarthritis

Exclusion Criteria:

* The patients with ASA score >II
* The patients with cancer
* The secondary coxarthrosis after the trauma
* Any vascular or neuromuscular diseases affecting the hip.

Ages: 70 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 80 (Actual)
Dates: Start 2006-05; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Stem migration in mm | 2 years

SECONDARY OUTCOMES:
Bone mineral density g/cm2 | 2 years
Temperature at bone-cement interface, degrees in Celsius | peroperatively
Serum- Titanium measurements in blood samples | Not defined

CONTACTS AND LOCATIONS:
Overall Officials: Mogens B Jørgensen, M.D., Principal Investigator — Northern Orthopaedic Division, Aalborg University Hospital, Denmark; Mogens B Laursen, M.D., Ph.D, Principal Investigator — Northern Orthopaedic Division, Aalborg University Hospital, Denmark; Lotte Borgwardt, dr., Principal Investigator — Frederikberg Hospital, Copenhagen; Kjeld Søballe, Ph.D., MD., Study Chair — University Hospital of Aarhus; Poul T Nielsen, M.D., Study Director — Northern Orthopaedic Division, Aalborg University Hospital, Denmark
Locations (1):
- Farsoe Hospital, Northern Orthopaedic Division, Farsø, Denmark